CLINICAL TRIAL: NCT03961035
Title: Comparative Effectiveness and Tolerance of Subliminal Subthreshold Transscleral Cyclophotocoagulation With a Duty Factor of 25 % Versus 31.3 % for Advanced Glaucoma
Brief Title: Comparative Effectiveness and Tolerance of Subliminal Subthreshold Transscleral Cyclophotocoagulation
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CPCTSI
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 25% cycle ratio: Patients group treated with CPCTSI at a 25% cycle ratio
- 31.3% cycle ratio: Patients group treated with CPCTSI at a 31.3% cycle ratio

SUMMARY:
Glaucoma, progressive optical neuropathy, is the leading cause of irreversible blindness in the world. Glaucoma treatment aims to lower intraocular pressure (IOP) by using medication, laser and surgery. Patients suffering from refractory and advanced glaucoma with impaired visual field who are not good candidates for surgery, cadenced subcleral transscleral cyclophotocoagulation (CPCTSI) is commonly used to reduce IOP. The CPCTSI consists in delivering short bursts of energy (in cycle) to the ciliary body, thus reducing production of aqueous humor. The energy gusts develop sequentially to a photocoagulating state in the pigmented epithelium. They are spaced by rest periods that allow surrounding tissue to cool down and remain below photocoagulative threshold, thus avoiding damage to surrounding tissue. Some studies have shown that the risk of complications increases with higher energies. Complications associated with CPCTSI include prolonged intraocular inflammation, pain, intraocular hemorrhage, hypotonia, phthysis, decreased vision and sympathetic ophthalmia. Severity of these complications depends on collateral damage inflicted on surrounding tissues: ciliary muscles, unpigmented epithelium and stroma of ciliary body. Currently, CPCTSI with a cycle ratio of 25% and 31.3% are used in surgical routine in ophthalmology. Cycle ratio is ratio between duration of gusts and total duration of cycle (gusts and rest periods). At St. Joseph's Hospital, both cycle ratios are used and the choice is operator dependent. However, using CPCTSI with a 25% cycle ratio could have fewer complications while maintaining similar efficacy. To our knowledge, there are no studies comparing these two cycle reports, although they are commonly used in practice. Our objective is to compare the CPCTSI with a cycle ratio of 25% and 31.3%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory and advanced glaucoma, defined as IOP > 21 mmHg according to maximum tolerated medical treatment, with or without pre-glaucoma surgical procedures and a visual field > 6 MD
* Patients treated in the GHPSJ ophthalmology department by a CPCTSI with cycle ratios of 25% or 31.3% between January and July 2017
* Patients who are poor candidates for additional filtration surgery or implantation of glaucoma drainage devices.

Exclusion Criteria:

* Patients who underwent intraocular surgery in the 2 months prior to CPCTSI
* Patients who have undergone conventional transscleral laser diode cyclophotocoagulation
* Patients who object to use of their data for this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory and advanced glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
Efficiency - Difference in success rates | Year 1
  Change in success rates between two groups of patients.

SECONDARY OUTCOMES:
Tolerance - Differences in occurrence frequency of side effects | Year 1
  Changes in occurrence frequency of side effects between two groups of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Yes